CLINICAL TRIAL: NCT00775138
Title: A Placebo Controlled, Randomized, Parallel Cohort, Safety And Tolerability Study Of 2 Dose Levels Of Liposomal Amikacin For Inhalation (Arikayce™) In Patients With Bronchiectasis Complicated By Chronic Infection Due To Pseudomonas Aeruginosa.
Brief Title: Safety and Tolerability Study of 2 Dose Level of Arikayce™ in Patients With Bronchiectasis and Chronic Infection Due to Pseudomonas Aeruginosa.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TR02-107
Record Dates: First submitted 2008-10-15; First posted 2008-10-17 (Estimated); Results first posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-06

CONDITIONS: Bronchiectasis
Keywords: Bronchiectasis; Respiratory Infections; Amikacin; Respiratory Tract Diseases; Respiratory Tract Infections; Lung Diseases; Pseudomonas aeruginosa; Amikacin liposome inhalation suspension (ALIS)
MeSH Terms: conditions — Bronchiectasis; Respiratory Tract Infections; Respiratory Tract Diseases; Lung Diseases; Pseudomonas Infections | interventions — Inhalation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 - 280 mg Arikayce™ (Experimental): Subjects in this arm of the cohort 1 will receive 280 mg of Arikayce™
  Interventions: Drug: 280 mg Arikayce™
- Cohort 1 - Placebo (Placebo Comparator): Subjects in this arm of the cohort 1 will receive matching placebo.
  Interventions: Drug: Matching Placebo for Cohort 1
- Cohort 2 - 560 mg Arikayce™ (Experimental): Subjects in this arm of the cohort 2 will receive 560 mg of Arikayce™
  Interventions: Drug: 560 mg Arikayce™
- Cohort 2 - Placebo (Placebo Comparator): Subjects in this arm of the cohort 2 will receive matching placebo
  Interventions: Drug: Matching Placebo for Cohort 2

INTERVENTIONS:
Drug: 280 mg Arikayce™ — Study subjects will receive Arikace™ 280 mg on Days 1 through Day 28. Drug is administered once a day via a nebulizer.
  Other Names: liposomal amikacin for inhalation
  Arms: Cohort 1 - 280 mg Arikayce™
Drug: Matching Placebo for Cohort 1 — Study subjects will receive placebo on Days 1 through Day 28. Drug is administered once a day via a nebulizer.
  Arms: Cohort 1 - Placebo
Drug: 560 mg Arikayce™ — Study subjects will receive Arikace™ 560 mg on Days 1 through Day 28. Drug is administered once a day via a nebulizer.
  Other Names: liposomal amikacin for inhalation
  Arms: Cohort 2 - 560 mg Arikayce™
Drug: Matching Placebo for Cohort 2 — Study subjects will receive placebo on Days 1 through Day 28. Drug is administered once a day via a nebulizer.
  Arms: Cohort 2 - Placebo

SUMMARY:
This is a study to determine the safety and tolerability of 28 days of daily dosing of two doses (280 mg and 560 mg) of Arikayce™ versus placebo in patients who have bronchiectasis and chronic infection due to Pseudomonas infection.

DETAILED DESCRIPTION:
Bronchiectasis is a chronic disorder of the major bronchi and bronchioles characterized by permanent dilation, microbial infection, a persistent inflammatory response with the release of immune mediators and microbial toxins leading to destruction. The origin of bronchiectasis varies, but the presence of microbial infection and a persistent inflammatory response is typical of the disease. The chronic nature of the infection and the associated considerable morbidity provides the rationale for using aerosolized antibiotics for the treatment of bronchiectasis patients.

This is a multi-national Phase 2 study of safety and tolerability of 28 days of daily dosing with two dose levels (280 mg and 560 mg) of Arikayce™ versus placebo in subjects with bronchiectasis and chronic Pseudomonas infection. Study subjects will be randomized to receive either study drug or placebo by inhalation via a PARI eFlow® nebulizer. Each subject will complete 28 days of daily dosing. All study subjects will be followed for microbiologic activity for 14 days after completion of treatment and for safety for 28 days post completion of study treatment.

The total study duration will be 56 days, with the screening visit occurring within the preceding 14 days prior to study day 1. At Day 1 (baseline), subjects will be evaluated at pre-dose and during the first 4-5 hours post-dose. Subjects will return at Week 2 (day 14) after start of treatment and at the end of Week 4 (Day 28) treatment period to determine safety and efficacy of Arikayce™. Subjects will be followed up on study Days 42 and 56 (about 2 and 4 weeks after end of treatment) for safety determination. After completion of this study, subjects will be followed up for an additional 6 months via phone contacts and records review, if hospitalized or treated for pulmonary exacerbation (under the extension protocol).

Clinical laboratory parameters, audiology testing, clinical adverse events and pulmonary function will be evaluated for all study subjects in order to determine the qualitative and quantitative safety and tolerability of Arikayce™ compared to placebo. Serum, urine and sputum specimens will be collected at periodic intervals to assess pharmacokinetics (PK) in subjects who consent for the PK portion of the study. Additionally, sputum samples will be collected to determine changes in bacterial density. Total Pulmonary Symptom Severity Score (PSSS) will be assessed, and respiratory quality of life will be evaluated by using the St. George's Respiratory Questionnaire (SGRQ). Arikace™,Arikayce™, Liposomal Amikacin for Inhalation (LAI), and Amikacin Liposome Inhalation Suspension (ALIS) may be used interchangeably throughout this study and the other studies evaluating amikacin liposome inhalation suspension.

ELIGIBILITY:
Inclusion Criteria:

* Male or female study subjects≥ 18 years of age
* Confirmed diagnosis of multi-focal bronchiectasis in two or more lung segments by HRCT of the chest
* History of chronic infection with P. aeruginosa
* Confirmation of infection with P. aeruginosa at screening
* SaO2 ≥ 90% at Screening while breathing room air
* Ability to comply with study medication use, study visits, and study procedures as judged by the investigator
* Ability to produce at least 0.5 grams sputum or be willing to undergo an induction to produce sputum for clinical evaluation

Key Exclusion Criteria:

* Forced Expiratory Volume in 1 second (FEV1) < 50% of predicted at Screening
* Patients with hemoptysis of ≥60 mL within 4 weeks prior to screening
* Bronchiectasis due to cystic fibrosis (CF), bronchopulmonary Aspergillus, aspiration of foreign body, or secondary to lung compression from tumors
* History of non-tuberculous mycobacterial and/or Aspergillus infection requiring treatment or treated within 2 years prior to screening
* Pulmonary tuberculosis requiring treatment or treated within two years prior to screening
* History of Lung transplantation
* Use of any inhalation or systemic antibiotics (IV antibiotics, or oral antibiotics) within 4 weeks prior to Study Day 1
* Evidence of biliary cirrhosis with portal hypertension
* Smoking tobacco or any substance within 6 months prior to screening, and throughout the study
* History of alcohol, medication, or illicit drug abuse within the 1 year prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-06-24 (Actual); Primary Completion 2009-05-11 (Actual); Study Completion 2009-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gina Eagle, MD, Study Director — Insmed Incorporated
Locations (18):
- United States (2):
  - Washington D.C., District of Columbia
  - Philadelphia, Pennsylvania
- Sofia, Bulgaria
- Athens, Greece
- Mosdós, Hungary
- India (6):
  - Bangalore
  - Hyderabad
  - Manipal
  - Mumbai
  - Nagpur
  - New Delhi
- Rabka-Zdrój, Poland
- Serbia (3):
  - Belgrade
  - Kragujevac
  - Niš
- Kiev, Ukraine
- United Kingdom (2):
  - Cambridge
  - London

RESULTS

PARTICIPANT FLOW:
Groups:
- Arikayce™ at 280 mg: Study subjects will receive Arikayce™ 280 mg on Days 1-28.
- Matching Placebo (280 mg); Matching Placebo (560 mg): Study subjects will receive matching placebo on Days 1-28.
- Arikayce™ at 560 mg: Study subjects will receive Arikayce™ 560 mg on Days 1-28.
Period: Overall Study
Arm/Group | Arikayce™ at 280 mg | Matching Placebo (280 mg) | Arikayce™ at 560 mg | Matching Placebo (560 mg)
Started | 24 | 10 | 20 | 10
Completed | 24 | 10 | 17 | 8
Not Completed | 0 | 0 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 2
Not completed — Adverse Event | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat (mITT) population, defined as all randomized patients who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arikayce™ at 280 mg | Matching Placebo (280 mg) | Arikayce™ at 560 mg | Matching Placebo (560 mg) | Total
Number analyzed (Participants) | 24 | 10 | 19 | 9 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (21.1) | 46.8 (15.0) | 58.5 (16.0) | 52.3 (11.1) | 52.4 (17.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 4 | 11 | 5 | 30
  Male | 14 | 6 | 8 | 4 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Treatment-emergent AEs (TEAEs) up to End of Treatment
Description: Number of Subjects reporting TEAE in the Arikayce™ groups and the placebo groups during the study. The table shows the events incidents, not the number of participants.
Time Frame: Day 1 through 56.
Population: Safety population, the same as the mITT population, defined as all randomized patients who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Arikace™ 280 mg: Study subjects will receive Arikace™ 280 mg on Days 1-28.
- Arikace™ 560 mg: Study subjects will receive Arikace™ 560 mg on Days 1-28.
Arm/Group | Arikace™ 280 mg | Matching Placebo (280 mg) | Arikace™ 560 mg | Matching Placebo (560 mg)
Number analyzed (Participants) | 24 | 10 | 19 | 9
Participants
  Productive Cough | 2 | 3 | 2 | 3
  Bronchial disorder | 3 | 0 | 1 | 0
  Cough | 1 | 2 | 5 | 0
  Haemoptysis | 2 | 1 | 1 | 0
  Pyrexia | 2 | 1 | 1 | 2
  Wheezing | 1 | 2 | 1 | 0
  Dyspnoea | 0 | 2 | 3 | 1
  Headache | 1 | 1 | 4 | 1
  Nasopharyngitis | 1 | 1 | 1 | 0
  Sneezing | 0 | 2 | 0 | 0
  Agitation | 1 | 0 | 0 | 0
  Aphthous stomatitis | 0 | 1 | 0 | 0
  Arthralgia | 1 | 0 | 0 | 0
  Cervicobrachial syndrome | 0 | 1 | 0 | 0
  Chronic obstructive pulmonary disease | 1 | 0 | 0 | 0
  Dizziness | 0 | 1 | 1 | 0
  Dysgeusia | 1 | 0 | 0 | 0
  Dysphonia | 1 | 0 | 2 | 0
  Forced expiratory volume decreased | 1 | 0 | 0 | 0
  Pharyngolaryngeal pain | 1 | 0 | 0 | 0
  Pruritus | 0 | 1 | 0 | 0
  Rash | 0 | 1 | 0 | 0
  Rhinorrhoea | 0 | 1 | 0 | 1
  Sinus bradycardia | 0 | 1 | 0 | 0
  Tinnitus | 1 | 0 | 0 | 0
  Toothache | 1 | 0 | 0 | 0
  Upper respiratory tract infection | 1 | 0 | 1 | 0
  Anorexia | 0 | 0 | 1 | 1
  Bronchiectasis | 0 | 0 | 1 | 1
  Fatigue | 0 | 0 | 1 | 1
  Insomnia | 0 | 0 | 1 | 1
  Abortion incomplete | 0 | 0 | 1 | 0
  Blood creatinine increased | 0 | 0 | 1 | 0
  Constipation | 0 | 0 | 0 | 1
  Laryngitis | 0 | 0 | 1 | 0
  Lung abscess | 0 | 0 | 0 | 1
  Nausea | 0 | 0 | 1 | 0
  Palpitations | 0 | 0 | 1 | 0

2. Primary Outcome: Treatment-emergent Marked Laboratory Abnormalities up to 28 Days After Study Medication Discontinuation
Description: Number of subjects reporting Incidence of clinically significant abnormalities in clinical values (Common Terminology Criteria for Adverse Events [CTCAE] grade >= 3) in Arikayce™ and placebo groups.
Time Frame: Day 1 through 56.
Population: The safety population is the mITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Arikace™ 280 mg | Matching Placebo (280 mg) | Arikace™ 560 mg | Matching Placebo (560 mg)
Number analyzed (Participants) | 24 | 10 | 19 | 9
Participants
  Leukocytes | 1 | 0 | 0 | 0
  Neutrophils Abs | 4 | 0 | 1 | 0
  Sodium | 1 | 0 | 0 | 0
  Uric acid | 0 | 1 | 1 | 1

3. Primary Outcome: Treatment-emergent Pulmonary Function Test (PFT) for Acute Tolerability Assessment
Description: Changes in PFT from pre-dose during the study were measured on Days 1, 14, and 28. Acute tolerability of the study treatment was assessed by examining the relative (rel.) changes in FEV1 from pre-dose assessments to 0-1 hour post-dose and 2-4 hours post-dose for each time point at which post-dose spirometry was conducted.
Time Frame: Pre-dose, 0-1 hour post-dose and 2-4 hours post-dose on day 1, 0-1 hour post-dose and 2-4 hours post-dose on day 14, and 0-1 hour post-dose and 2-4 hours post-dose on day 28
Population: The analysis population is the safety population, the same as the mITT population, defined as all randomized patients who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Arikace™ 280 mg | Matching Placebo (280 mg) | Arikace™ 560 mg | Matching Placebo (560 mg)
Number analyzed (Participants) | 24 | 10 | 19 | 9
L
  Day 1: Pre-Dose | 1.917 (0.793) | 1.841 (0.536) | 1.939 (0.515) | 1.758 (0.654)
  Day 1: 0 - 1 Hr Post-Dose | 1.922 (0.780) | 1.820 (0.546) | 1.907 (0.475) | 1.807 (0.666)
  Day 1: 2 - 4 Hrs Post-Dose | 1.955 (0.766) | 1.864 (0.520) | 1.912 (0.477) | 1.812 (0.675)
  Day1:0-1 Hr Post-Dose Rel. Change from Pre-dose | 0.816 (9.317) | -1.186 (3.028) | -0.873 (9.640) | 3.128 (12.088)
  Day1:2-4 Hrs Post-Dose Rel. Change from Pre-dose | 3.323 (11.181) | 1.484 (3.507) | -0.661 (8.374) | 3.082 (11.671)
  Day 14: Pre-Dose | 1.892 (0.759) | 1.761 (0.550) | 1.864 (0.607) | 1.895 (0.592)
  Day 14: 0 - 1 Hr Post-Dose | 1.907 (0.776) | 1.794 (0.556) | 1.856 (0.555) | 1.908 (0.611)
  Day 14: 2 - 4 Hr Post-Dose | 1.931 (0.771) | 1.797 (0.520) | 1.843 (0.567) | 1.901 (0.542)
  Day14:0-1 Hr Post-Dose Rel. Change from Pre-dose | 0.800 (8.818) | 2.061 (4.509) | -1.629 (9.961) | 0.589 (4.558)
  Day14:2-4 Hr Post-Dose Rel. Change from Pre-dose | 2.388 (9.020) | 2.711 (6.620) | -3.114 (8.506) | 1.228 (9.617)
  Day 28: Pre-Dose | 1.919 (0.761) | 1.794 (0.507) | 1.846 (0.532) | 1.934 (0.560)
  Day 28: 0 - 1 Hr Post-Dose | 1.928 (0.751) | 1.803 (0.502) | 1.797 (0.541) | 1.901 (0.550)
  Day 28: 2 - 4 Hrs Post-Dose | 1.908 (0.754) | 1.809 (0.527) | 1.799 (0.578) | 1.940 (0.641)
  Day 28:0-1 Hr Post-Dose Rel. Change from Pre-dose | 0.635 (7.647) | 0.654 (3.675) | 0.607 (4.185) | -1.437 (6.454)
  Day 28:2-4 Hrs Post-Dose Rel. Change from Pre-dose | -0.356 (8.858) | 0.601 (3.184) | -0.006 (6.156) | -0.542 (7.690)

4. Primary Outcome: Treatment-emergent PFT Abnormalities up to the End of Study
Description: Number of Subjects with Decrease of >= 15% in FEV1 (L) from Pre- to Post-dose by Study Day
Time Frame: Day 1, Day 14 and Day 28
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Arikace™ 280 mg | Matching Placebo (280 mg) | Arikace™ 560 mg | Matching Placebo (560 mg)
Number analyzed (Participants) | 24 | 10 | 19 | 9
Participants
  Day 1: No | 22 | 10 | 17 | 9
  Day 1: Yes | 2 | 0 | 2 | 0
  Day 14: No | 23 | 10 | 18 | 9
  Day 14: Yes | 1 | 0 | 1 | 0
  Day 28: No | 23 | 10 | 19 | 9
  Day 28: Yes | 1 | 0 | 0 | 0

5. Primary Outcome: Number of Subjects With an Adverse Event Leading to Permanent Discontinuation of Study Medication
Time Frame: Screening to Day 56
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Arikace™ 280 mg | Matching Placebo (280 mg) | Arikace™ 560 mg | Matching Placebo (560 mg)
Number analyzed (Participants) | 24 | 10 | 19 | 9
Participants | 0 | 0 | 1 | 0

6. Primary Outcome: Serious Adverse Events up to 28 Days After Study Medication Discontinuation
Description: Number of subjects with a SAE in the Arikace™ groups and the placebo group up to 28 days after study medication discontinuation. See SAE table in the safety section for details.
Time Frame: Screening to Day 56
Population: The safety population is the modified intent-to-treat (mITT) population, defined as all randomized patients who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Arikace™ 560 mg: Study subjects will receive Arikace™ 280 mg on Days 1-28.
Arm/Group | Arikace™ 280 mg | Matching Placebo (280 mg) | Arikace™ 560 mg | Matching Placebo (560 mg)
Number analyzed (Participants) | 24 | 10 | 19 | 9
Participants | 1 | 0 | 1 | 1

7. Secondary Outcome: Change From Baseline in Log10CFU Per Gram (Density) of Pseudomonas Aeruginosa in Sputum.
Description: The change in Pseudomonas aeruginosa density from from baseline to Day 14, 28, and 42 were evaluated.Treatment differences with respect to the changes from baseline to each measured study day, defined as the log10 of the sum of all morphotypes (colony-forming units [CFU]) per gram of sputum in (log10CFU/gram [g]), was estimated for each treatment group; standard deviations accompanied the treatment differences.
Time Frame: Baseline to Day 14, Day 28 and Day 42.
Population: Per source, this is the Pa population, which includes patients who grew Pa on day 1, analyzed as treated.
Measure: Mean (Standard Deviation); unit: log10CFU per gram
Arm/Group | Arikace™ 280 mg | Matching Placebo (280 mg) | Arikace™ 560 mg | Matching Placebo (560 mg)
Number analyzed (Participants) | 17 | 9 | 15 | 8
log10CFU per gram
  Day 14 Change from Baseline | -0.227 (0.805) | -0.333 (0.515) | -2.016 (1.942) | -0.474 (1.942)
  Day 28 Change from Baseline | -0.094 (0.975) | 0.315 (0.732) | -1.013 (1.099) | -0.302 (0.443)
  Day 42 Change from Baseline | 0.101 (0.788) | -0.057 (0.627) | 0.046 (0.705) | -0.641 (1.095)

8. Secondary Outcome: Total Pulmonary Symptom Severity Score (PSSS)
Description: Changes in the severity and intensity (frequency x severity) of individual symptoms and change in composite PSSS from baseline to Days 14, 28, 42 and 56.
  The Pulmonary Symptom Severity Score (PSSS) was assessed on patient's responses to the Patients Symptoms Questionnaire, which employs symptom frequency and severity scales described for the validated Memorial Symptoms Assessment Scale. Symptom severity was scored on a scale of 0 (not applicable or symptom not present) to 4 (very severe) for each of the 5 symptoms (cough, shortness of breath, sputum production [frequency and severity], fatigue, and wheezing), and a composite score (range, 0 to 20 [low score represents better outcome]) was obtained as the sum of the severity scores for each symptom.
Time Frame: Baseline to Day 14, Day 28, Day 42 and Day 56.
Population: The safety population is used for this analysis. It is the same as the mITT population, defined as all randomized patients who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arikace™ 280 mg | Matching Placebo (280 mg) | Arikace™ 560 mg | Matching Placebo (560 mg)
Number analyzed (Participants) | 24 | 10 | 19 | 9
score on a scale
  Day 14 change from Day 1 | -1.125 (2.213) | -0.200 (0.789) | -0.471 (2.035) | -0.250 (2.053)
  Day 28 change from Day 1 | -2.167 (2.988) | 0.000 (2.357) | -1.000 (4.087) | -0.125 (4.257)
  Day 42 change from Day 1 | -2.458 (3.476) | -1.000 (1.491) | -1.882 (4.285) | 1.125 (3.137)
  Day 56 change from Day 1 | -2.458 (2.874) | -1.500 (2.121) | -2.167 (3.053) | -2.000 (1.690)

9. Secondary Outcome: To Evaluate Change in St. George's Respiratory Questionnaire Measurements
Description: A composite total score is derived as the sum of domain scores for symptoms, activity, and impact, with 0 as the best possible score and 100 as the worst possible score. A reduction in score of 4 points is generally recognized as a clinically meaningful improvement in quality of life. This analysis compared the changes from Day 1 (prior to first dosing) to Days 14, 28, 42, and 56.
Time Frame: Day 1 to Day 14, Day 28, Day 42 and Day 56.
Population: The analysis population is the mITT population, defined as all randomized patients who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arikace™ 280 mg | Matching Placebo (280 mg) | Arikace™ 560 mg | Matching Placebo (560 mg)
Number analyzed (Participants) | 24 | 10 | 19 | 9
score on a scale
  Day 14 change from Day 1 | -4.024 (8.558) | -6.350 (8.756) | -6.101 (12.164) | -2.807 (7.256)
  Day 28 change from Day 1 | -6.205 (13.661) | -5.812 (12.039) | -6.200 (11.855) | -8.304 (12.993)
  Day 42 change from Day 1 | -7.611 (13.274) | -6.130 (14.271) | -8.196 (12.332) | 0.242 (5.818)
  Day 56 change from Day 1 | -7.937 (16.281) | -7.371 (11.270) | -9.282 (10.302) | -1.637 (15.161)

10. Secondary Outcome: To Evaluate the Use of Systemic Antipseudomonal Rescue Therapy
Time Frame: Screening to Day 56.
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Groups:
- Matching Placebo (280mg); Matching Placebo (560 mg): Study subjects will receive matching placebo on Days 1-28.
Arm/Group | Arikace™ 280 mg | Matching Placebo (280mg) | Arikace™ 560 mg | Matching Placebo (560 mg)
Number analyzed (Participants) | 24 | 10 | 19 | 9
Participants
  Rescue Medication Initiation by Day 28 | 0 | 0 | 0 | 1
  Rescue Medication Initiation by Day 56 | 0 | 0 | 0 | 1
  No Rescue Medication Initiation | 24 | 10 | 19 | 7

ADVERSE EVENTS:
Time Frame: TEAEs were assessed at Baseline and all subsequent study visits up to day 56
Groups:
- Arikace at 280 mg: Study subjects will receive Arikace™ 280 mg on Days 1-28.
- Arikace at 560 mg: Study subjects will receive Arikace™ 560 mg on Days 1-28.
Arm/Group | Arikace at 280 mg | Matching Placebo (280 mg) | Arikace at 560 mg | Matching Placebo (560 mg)
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/10 | 0/19 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/24 | 0/10 | 1/19 | 1/9
Other Adverse Events (participants affected / at risk) | 11/24 | 5/10 | 11/19 | 6/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arikace at 280 mg (N=24) | Matching Placebo (280 mg) (N=10) | Arikace at 560 mg (N=19) | Matching Placebo (560 mg) (N=9)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion Incomplete (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung Abscess (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arikace at 280 mg (N=24) | Matching Placebo (280 mg) (N=10) | Arikace at 560 mg (N=19) | Matching Placebo (560 mg) (N=9)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aphthous Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (3)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Bronchiectasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Creatinine Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heart Rate Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (3) | 4 (4) | 1 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (21) | 1 (1) | 0 (0)
Cervicobrachial Syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4) | 2 (3) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (4) | 5 (11) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 3 (3) | 1 (1)
Bronchial Disorder (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes